CLINICAL TRIAL: NCT03897829
Title: Prevalence of Knee Cap Enthesitis in Patients With Knee Osteoarthritis, Cross Sectional Ultrasonographic Study.
Brief Title: Enthesitis in Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Abogamal, Professor, Al-Azhar University
Other Study IDs: aswu/320/1/19
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Osteoarthritis
Keywords: enthesitis; osteoarthritis; ultrasound
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current study was conducted to estimate the prevalence of knee cap enthesitis in patients with knee osteoarthritis and its relation to knee function.

DETAILED DESCRIPTION:
The current study will based on a cross sectional hospital-based survey, conducted among patients with knee osteoarthritis , Knee will assessed for the following items in both sides while Patient lying supine with the knee flexed 40 degrees:

1. Superior pole of the patella - quadriceps tendon enthesis: ● Quadriceps tendon thickness >6.1 mm ● Suprapatellar bursitis ● Superior pole of patella erosion ● Superior pole of patella enthesophyte.
2. Inferior pole of the patella - proximal patellar ligament enthesis: ● Patellar ligament thickness >4 mm ● Inferior pole of patella erosion ● Inferior pole of patella enthesophyte.
3. Tibial tuberosity - distal patellar ligament enthesis ● Patellar ligament thickness >4 mm ● Infrapatellar bursitis ● Tibial tuberosity erosion ● Tibial tuberosity enthesophyte.

Knee functional status was assessed using Knee injury and Osteoarthritis Outcome Score (KOOS) scale for Pain, other Symptoms, Activities of Daily Living (ADL), Sport and Recreation Function (Sport/Rec) and knee-related Quality of Life (QOL). Low knee function was considered if the patient had score 50 or more in any KOOS scale parameter.

ELIGIBILITY:
Inclusion Criteria:

* Primary Knee OA diagnosed according to: American College of Rheumatology Radiologic Criteria for Knee Osteoarthritis.
* Kellegren - Lawrance scale grade II.
* On regular treatment by analgesics, or NSAIDS either topical or systemic.

Exclusion Criteria:

* Recent Knee trauma or intra-articular procedures.
* Previous knee surgery.
* Inflammatory joint diseases, as rheumatoid arthritis, crystal arthritis, and spondyloarthropathy
* chronic systemic diseases that could affect patient functional ability; e.g renal, liver, cardiac impairment, or neurological disorder.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The current study will be based on a cross-sectional hospital-based survey, conducted among patients with knee osteoarthritis presenting at outpatient rheumatology clinics of AL-AZHAR University Hospitals, and Aswan university hospital according to the inclusion-exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of knee cap enthesitis in patients with knee osteoarthritis | two months
  Detection of the prevalence

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Al-Azhar Faculty of medicine, Rheumatology Department, Cairo
  - Al-Azhar university hospitals, Cairo

IPD SHARING:
Plan to Share IPD: Undecided
not yet decided